CLINICAL TRIAL: NCT01792440
Title: The Sputum Colour Chart as a Predictor of Lung Inflammation, Proteolysis and Damage in Non-cystic Fibrosis Bronchiectasis
Brief Title: The Sputum Colour Chart as a Predictor of Lung Inflammation and Proteolysis in Non-cystic Fibrosis Bronchiectasis
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Dr. Lieven Dupont, prof. dr., Universitaire Ziekenhuizen KU Leuven
Other Study IDs: B32220084152; B51060 (Other: Belgium: Institutional Review Board)
Record Dates: First submitted 2013-02-13; First posted 2013-02-15 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Non-cystic Fibrosis Bronchiectasis; Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — induced sputum cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- non-cystic fibrosis bronchiectasis: patients with non-cystic fibrosis bronchiectasis will be evaluated cross-sectionally
- healthy control subjects: healthy control subjects will be evaluated cross-sectionally

SUMMARY:
Non-cystic fibrosis bronchiectasis patients (and controls) were recruited for the study. The investigators' aim was to study the relevance of clinical parameters in terms of underlying disease severity, proteolysis and inflammation in a diverse non-cystic fibrosis bronchiectasis population.

DETAILED DESCRIPTION:
Patients from the non-cystic fibrosis bronchiectasis (NCFB) outpatient clinic were recruited in our study from September 2009 till July 2010. Control healthy subjects were recruited among peers of the patient or hospital staff during the same period. For the NCFB patients, underlying etiologies of NCFB and Pseudomonas aeruginosa (PA) colonization status were analyzed and each patient was evaluated by means of spirometry (FVC and FEV1), Leicester Cough Questionnaire (LCQ) and Sputum Colour Chart (SCC). SCC assessment was both done by letting the patient predict his sputum purulence prior to sputum induction and by SCC scoring after sputum harvest by the physician.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of NCFB, based on CT findings of bronchiectatic disease in the absence of cystic fibrosis (CF) as a cause.
* stable

Exclusion Criteria:

* no recent exacerbation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: non-cystic fibrosis bronchiectasis
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2009-09; Primary Completion 2010-07 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Assess predictive value of sputum colour chart to evaluate airway inflammation | 10 months
  Airway inflammation will be assessed by analysis of sputum differential cell counts and cytokine/chemokine analysis in sputum.

SECONDARY OUTCOMES:
Link the degree of airway inflammation to the proteolytic activity of sputum enzymes. | 10 months
  Proteolytic activity of sputum enzymes (total gelatinolytic activity) and sputum enzymes (neutrophil elastase, MMP9) will be quantified in sputum supernatant of NCFB patients and controls.

CONTACTS AND LOCATIONS:
Overall Officials: Pieter Goeminne, MD, Study Director — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospital Leuven, Leuven, Vlaams-Brabent, Belgium